CLINICAL TRIAL: NCT00803738
Title: A Multi-center, Randomized, Investigator-blinded, Parallel-group Study, Designed to Evaluate the Safety and Clinical Equivalence of Terconazole Vaginal Suppositories, 80 mg (Test Product) and Terconazole Vaginal Suppositories, 80 mg (Reference Product) in the Treatment of Vulvovaginal Candidiasis Caused by Candida Species
Brief Title: Safety and Equivalence of a Terconazole Vaginal Suppository (Test Product) Compared to the Reference Terconazole Vaginal Suppository in the Treatment of Vulvovaginal Candidiasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Padagis LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CPL-202
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Results first posted 2013-02-20 (Estimated); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Vulvovaginal Candidiasis
Keywords: Vulvovaginal Candidiasis; Terconazole
MeSH Terms: conditions — Candidiasis, Vulvovaginal

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test Product (Experimental): Terconazole Vaginal Suppository
  Interventions: Drug: Terconazole Vaginal Suppository
- Reference Product (Active Comparator): Terazol Vaginal Suppository
  Interventions: Drug: Terazol Vaginal Suppository

INTERVENTIONS:
Drug: Terconazole Vaginal Suppository — Vaginal Suppository inserted intravaginally once daily before bedtime for 3 consecutive days
  Arms: Test Product
Drug: Terazol Vaginal Suppository — Vaginal Suppository inserted intravaginally once daily before bedtime for 3 consecutive days
  Other Names: Terazol 3 suppository
  Arms: Reference Product

SUMMARY:
The objectives of this study were to demonstrate comparable safety and efficacy of Terconazole Vaginal Suppositories, 80 mg(Test Product) and Terconazole Vaginal Suppositories, 80 mg(Reference Product) in the treatment of subjects with vulvovaginal candidiasis in order to establish bioequivalence.

ELIGIBILITY:
Inclusion Criteria:

* Female at least 18 years of age
* Presented with symptomatic vulvovaginitis consistent with a diagnosis of moniliasis
* Willing and able to read and sign an IRB approved ICF, which included agreement to comply with all study requirements as indicated in the protocol.

Exclusion Criteria:

* History of hypersensitivity or allergy to imidazoles
* Female who was pregnant or lactating
* Was menstruating or expected the onset of menses during the treatment days
* Had evidence of any bacterial, viral or protozoal infection
* Had a history of alcoholism, drug abuse, or problems that would likely have made the subject unreliable for the study
* Had any condition or used any medication that, in the opinion of the Investigator, might have interfered with the conduct or results of the study or placed the prospective subject at increased risk
* Had participated in any investigational study within 30 days prior to study enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 572 (Actual)
Dates: Start 2002-12; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at 31 dermatology clinical practices.
Groups:
- Terconazole Vaginal Suppositories, 80 mg - Perrigo: Terconazole Vaginal Suppositories, 80 mg manufactured by Perrigo applied intravaginally once daily before bedtime for 3 consecutive days
- Terazol 3 - Terconazole Vaginal Suppositories 80 mg: Terazol 3 manufactured by Ortho-McNeil Pharmaceutical, Inc applied intravaginally once daily before bedtime for 3 consecutive daysapplied the study medication intravaginally once daily before bedtime for 3 consecutive days
Period: Overall Study
Arm/Group | Terconazole Vaginal Suppositories, 80 mg - Perrigo | Terazol 3 - Terconazole Vaginal Suppositories 80 mg
Started | 286 | 286
Completed | 192 | 176
Not Completed | 94 | 110
Not completed — Adverse Event | 3 | 5
Not completed — Lost to Follow-up | 4 | 4
Not completed — Protocol Violation | 18 | 10
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Lack of Efficacy | 10 | 16
Not completed — Negative Baseline Culture of Candida | 56 | 63
Not completed — Positive Results for STD or abnormal PAP | 2 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Terconazole Vaginal Suppositories, 80 mg - Perrigo | Terazol 3 - Terconazole Vaginal Suppositories 80 mg | Total
Number analyzed (Participants) | 286 | 286 | 572
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 278 | 276 | 554
  >=65 years | 8 | 10 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.4 (13.3) | 31.6 (13.1) | 32.5 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 286 | 286 | 572
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 286 | 286 | 572

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects in Each Treatment Group With Therapeutic Cure
Description: The primary efficacy measure was the proportion of subjects in each treatment group with a therapeutic cure at the Test-of-Cure visit (Visit 3). A subject was considered a therapeutic cure if the subject was a clinical cure with mycological cure.
Time Frame: Visit 3: Day 22-31
Population: Per Protocol (PP) population
Measure: Number; unit: participants
Arm/Group | Terconazole Vaginal Suppositories, 80 mg - Perrigo | Terazol 3 - Terconazole Vaginal Suppositories 80 mg
Number analyzed (Participants) | 153 | 147
participants | 105 [-4.3 to 15.02] | 93 [-4.3 to 15.02]
Statistical Analysis 1: Comparison: Terconazole Vaginal Suppositories, 80 mg - Perrigo vs Terazol 3 - Terconazole Vaginal Suppositories 80 mg; Test type: Non-Inferiority or Equivalence — For the primary clinical equivalence analysis, a 90% confidence interval was constructed on the difference in the therapeutic cure rates between the Test Product and Reference Product at the Test-of-Cure visit (Visit 3). The interval was calculated using Wald's method with Yates' continuity correction. Clinical equivalence was established if this 90% confidence interval was contained within the interval -0.20 to +0.20 (-20% to +20%); Wald's method with Yates' continuity; proportion of subjects in trtmt groups = .05, 90% CI 2-sided [-4.30 to 15.02]

2. Secondary Outcome: Proportion of Subjects With Mycological Cure
Description: Mycological cure was defined as a negative mycological culture (no growth) for Candida albicans or other relevant baseline yeast organism.
Time Frame: Visit 3: Day 22-31
Population: Per protocol population
Measure: Number; unit: participants
Arm/Group | Terconazole Vaginal Suppositories, 80 mg - Perrigo | Terazol 3 - Terconazole Vaginal Suppositories 80 mg
Number analyzed (Participants) | 153 | 147
participants | 127 | 117
Statistical Analysis 1: Comparison: Terconazole Vaginal Suppositories, 80 mg - Perrigo vs Terazol 3 - Terconazole Vaginal Suppositories 80 mg; Test type: Non-Inferiority or Equivalence — A 90% confidence interval was constructed on the difference in the mycological cure rates between the Test Product and Reference Product at the Test-of-Cure visit (Visit 3). The interval was calculated using Wald's method with Yates' continuity correction. Clinical equivalence was established if this 90% confidence interval was contained within the interval -0.20 to +0.20 (-20% to +20%); Wald's method with Yates' continuity; proportion of subjects in trtmt groups = .05, 90% CI 2-sided [-4.66 to 11.49]

3. Secondary Outcome: Proportion of Subjects With Clinical Cure
Description: A subject was considered a clinical cure if all of the following were satisfied:
  1. All signs and symptoms with a score of 1 (mild) or 2 (moderate) at the Screening/Baseline visit were absent (score = 0), and all signs or symptoms with a score of 3 (severe) at Screening/Baseline had a score of 0 or 1.
  2. Total signs and symptoms did not worsen at any time following completion of the study treatment.
  3. Any new sign or symptom observed during the study period was determined by the Investigator not to be related to VVC.
  4. The subject did not require additional vulvovaginal or systemic antifungal therapy at any time during the study period.
  5. The subject did not use any topical drug therapy other than the study medication for the treatment of vulvovaginal irritation and/or pruritus such as topical analgesic or corticosteroid products
Time Frame: Visit 3: Day 22-31
Population: per protocol population
Measure: Number; unit: participants
Arm/Group | Terconazole Vaginal Suppositories, 80 mg - Perrigo | Terazol 3 - Terconazole Vaginal Suppositories 80 mg
Number analyzed (Participants) | 153 | 147
participants | 117 | 101
Statistical Analysis 1: Comparison: Terconazole Vaginal Suppositories, 80 mg - Perrigo vs Terazol 3 - Terconazole Vaginal Suppositories 80 mg; Test type: Non-Inferiority or Equivalence — A 90% confidence interval was constructed on the difference in the clinical cure rates between the Test Product and Reference Product at the Test-of-Cure visit (Visit 3). The interval was calculated using Wald's method with Yates' continuity correction. Clinical equivalence was established if this 90% confidence interval was contained within the interval -0.20 to +0.20 (-20% to +20%); Wald's method with Yates' continuity; proportion of subjects in trtmt groups = .05, 90% CI 2-sided [-1.35 to 16.88]

ADVERSE EVENTS:
Time Frame: Up to day 31
Description: Incidence of AEs during the study was summarized by treatment group. Frequency of all AEs was tabulated by treatment group, COSTART body system, severity, and relationship to the study medication. The differences between the treatment groups were compared using statistical measures. The analyses were conducted in the ITT population only.
Arm/Group | Terconazole Vaginal Suppositories, 80 mg - Perrigo | Terazol 3 - Terconazole Vaginal Suppositories 80 mg
Serious Adverse Events (participants affected / at risk) | 0/282 | 1/275
Other Adverse Events (participants affected / at risk) | 48/282 | 54/275
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Terconazole Vaginal Suppositories, 80 mg - Perrigo (N=282) | Terazol 3 - Terconazole Vaginal Suppositories 80 mg (N=275)
appendicitis (Infections and infestations) | 0 (0) | 1 (1) — The event met the criteria for an SAE. The SAE was considered by the investigator to be unrelated to study medication. The subject completed the study and was included in the MITT analyses
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Terconazole Vaginal Suppositories, 80 mg - Perrigo (N=282) | Terazol 3 - Terconazole Vaginal Suppositories 80 mg (N=275)
headache (Nervous system disorders) | 36 (36) | 39 (39)
infection (Infections and infestations) | 12 (12) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other